CLINICAL TRIAL: NCT02796677
Title: A 24 Week Treatment, Multicenter, Randomized, Double Blinded, Double Dummy, Parallel-group, Clinical Trial Evaluating the Efficacy and Safety of Aclidinium Bromide 400 μg/Formoterol Fumarate 12 μg Fixed-dose Combination BID Compared With Each Monotherapy (Aclidinium Bromide 400 μg BID and Formoterol Fumarate 12 μg BID) and Tiotropium 18 μg QD When Administered to Patients With Stable Chronic Obstructive Pulmonary Disease.
Brief Title: AMPLIFY - D6571C00001 Duaklir USA Phase III Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6571C00001
Record Dates: First submitted 2016-05-31; First posted 2016-06-13 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Safety; Efficacy; Aclidinium bromide; Formoterol fumarate; Tiotropium; Bronchodilation; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide; Formoterol Fumarate; Inhalation; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- AB/FF 400/12 μg BID (Experimental): Participants were administered AB/FF 400/12 μg via Pressair®/Genuair® inhaler twice daily for 24 weeks of treatment.
  Interventions: Drug: Aclidinium bromide 400 μg/Formoterol Fumarate 12 μg (AB/FF 400/12 μg); Other: Placebo to AB/FF 400/12 μg, AB 400 μg and FF 12 μg
- AB 400 μg BID (Experimental): Participants were administered AB 400 μg via Pressair®/Genuair® inhaler twice daily for 24 weeks of treatment.
  Interventions: Drug: Aclidinium bromide 400 μg (AB 400 μg); Other: Placebo to AB/FF 400/12 μg, AB 400 μg and FF 12 μg
- FF 12 μg BID (Experimental): Participants were administered FF 12 μg via Pressair®/Genuair® inhaler twice daily for 24 weeks of treatment.
  Interventions: Drug: Formoterol fumarate 12 μg (FF 12 μg); Other: Placebo to AB/FF 400/12 μg, AB 400 μg and FF 12 μg
- TIO 18 μg QD (Experimental): Participants were administered TIO 18 μg via Handihaler® inhale once daily for 24 weeks of treatment.
  Interventions: Drug: Tiotropium 18 μg (TIO 18 μg); Other: Placebo to TIO 18 μg

INTERVENTIONS:
Drug: Aclidinium bromide 400 μg/Formoterol Fumarate 12 μg (AB/FF 400/12 μg) — Inhalation powder
  Other Names: Oral Inhalation (by Pressair®/Genuair® Dry Powder Inhaler)
  Arms: AB/FF 400/12 μg BID
Drug: Aclidinium bromide 400 μg (AB 400 μg) — Inhalation powder
  Other Names: Oral Inhalation (by Pressair®/Genuair® Dry Powder Inhaler)
  Arms: AB 400 μg BID
Drug: Formoterol fumarate 12 μg (FF 12 μg) — Inhalation powder
  Other Names: Oral Inhalation (by Pressair®/Genuair® Dry Powder Inhaler)
  Arms: FF 12 μg BID
Other: Placebo to AB/FF 400/12 μg, AB 400 μg and FF 12 μg — Inhalation powder
  Other Names: Oral Inhalation (by Pressair®/Genuair® Dry Powder Inhaler)
  Arms: AB 400 μg BID; AB/FF 400/12 μg BID; FF 12 μg BID
Drug: Tiotropium 18 μg (TIO 18 μg) — Powder in capsules for oral inhalation
  Other Names: Oral Inhalation (by Handihaler® Dry Powder Inhaler, DPI)
  Arms: TIO 18 μg QD
Other: Placebo to TIO 18 μg — Powder in capsules for oral inhalation
  Other Names: Oral Inhalation (by Handihaler® Dry Powder Inhaler, DPI)
  Arms: TIO 18 μg QD

SUMMARY:
This is a multiple dose, randomized, parallel, double-blind, double-dummy, multicenter and multinational Phase III study to determine the efficacy and safety of Aclidinium bromide 400μg/Formoterol Fumarate (AB/FF) 12 μg compared to individual components and TIO (Tiotropium) 18 μg when administered to patients with stable chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
This study was conducted to assess the bronchodilator efficacy and safety as well as effect on health related quality of life of AB/FF 400/12 μg compared to the individual components (AB 400 μg and FF 12 μg) in COPD patients. The trial duration of 24 weeks allows the assessment of the effect on symptoms improvement of the combined treatments versus individual components as well as the long term bronchodilation comparison between AB 400 μg and TIO 18 μg in minimizing the risk of COPD exacerbations in current or former smokers, aged ≥40 in symptomatic COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or non-pregnant, non-lactating female patients aged ≥40.
* Patients with diagnosis of moderate to very severe stable COPD: post-bronchodilator FEV1 < 80% of the predicted normal and post-bronchodilator FEV1/FVC < 70% at Screening Visit.
* Symptomatic patients with a CAT score ≥10 at Screening and Randomization visit (Visits 1 and 2).
* Current or former-smokers, with a smoking history of ≥ 10 pack-years.
* Patients able to perform acceptable and repeatable pulmonary function testing for FEV1 according to the American Thoracic Society (ATS)/European Respiratory Society (ERS) 2005 criteria at Visit 1.
* Patients eligible and able to participate in the study and who had signed an Informed Consent Form prior to initiation of any study-related procedures.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to AstraZeneca staff and/or site staff), or patients employed by or relatives of the employees of the site or sponsor.
* Previous randomization in the present study D6571C00001.
* Patients with predominant asthma.
* Any respiratory tract infection (including the upper respiratory tract) or COPD exacerbation (including the mild COPD exacerbation) within 6 weeks prior to screening or during the run-in period.
* Patients hospitalized for a COPD exacerbation (an emergency room visit for longer than 24 hours is considered a hospitalization) within 3 months prior to Screening Visit.
* Clinically significant respiratory conditions other than COPD.
* Patients who in the Investigator's opinion may need to start a pulmonary rehabilitation program during the study and/or patients who started/finished it within 3 months prior to Screening.
* Use of long-term oxygen therapy (≥ 15 hours/day).
* Patients who do not maintain regular day/night, waking/sleeping cycles including night shift workers.
* Clinically significant cardiovascular conditions.
* Patients with uncontrolled Type I or Type II diabetes, uncontrolled hypo-or hyperthyroidism, hypokalaemia, or hyperadrenergic state, uncontrolled hypertension.
* Patients with history of long QT syndrome or whose QTc (calculated according to Fridericia's Formula QTc=QT/RR1/3) > 470 ms as indicated in the centralised reading report assessed at Screening.
* Patients with clinically significant abnormalities in the laboratory tests, ECG parameters (other than QTc) or in the physical examination at Screening Visit that might comprise patient safety.
* Patient with known non-controlled history of infection with human immunodeficiency virus and/or active hepatitis.
* Patient with a history of hypersensitivity reaction to inhaled medication or any component thereof, including paradoxical bronchospasm.
* Patients with known narrow-angle glaucoma, symptomatic bladder neck obstruction, acute urinary retention or symptomatic non-stable prostate hypertrophy.
* History of malignancy of any organ system (including lung cancer), treated or untreated, within the past 5 years other than basal or squamous cell skin cancer.
* Patients with any other serious or uncontrolled physical or mental dysfunction.
* Patients with a history (within 2 years prior to screening) of drug and/or alcohol abuse that may prevent study compliance based on the Investigator judgment.
* Patients unlikely to be cooperative or that cannot comply with the study procedures.
* Patients treated with any investigational drug within 30 days (or 6 half-lives, whichever is longer) prior to Screening.
* Patients who intended to use any concomitant medication not permitted by this protocol or who had not undergone the required washout period for a particular prohibited medication.
* Patients unable to give consent, or patients of consenting age but under guardianship, or vulnerable patients. Patients who demonstrate < 80% compliance with the electronic diary during the run-in period.

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1595 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Sethi, Principal Investigator — 3495 Bailey Ave , Buffalo NY14215, USA
Locations (146):
- United States (77):
  - Research Site, Gulf Shores, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Corona, California
  - Research Site, Fresno, California
  - Research Site, Fullerton, California
  - Research Site, Lincoln, California
  - Research Site, San Diego, California
  - Research Site, Waterbury, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Edgewater, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Homestead, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Blue Ridge, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Portage, Indiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Fall River, Massachusetts
  - Research Site, Chelsea, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, Fridley, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Woodbury, Minnesota
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Fremont, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Grove City, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Midwest City, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Columbia, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Union, South Carolina
  - Research Site, Arlington, Texas
  - Research Site, Baytown, Texas
  - Research Site, Boerne, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Lewisville, Texas
  - Research Site, McKinney, Texas
  - Research Site, Tomball, Texas
  - Research Site, Midvale, Utah
  - Research Site, Abingdon, Virginia
  - Research Site, Newport News, Virginia
- Bulgaria (9):
  - Research Site, Dimitrovgrad
  - Research Site, Gabrovo
  - Research Site, Roman
  - Research Site, Rousse
  - Research Site, Sevlievo
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Vidin
- Czechia (5):
  - Research Site, Jaroměř
  - Research Site, Jindřichův Hradec
  - Research Site, Prague
  - Research Site, Rokycany
  - Research Site, Strakonice
- Germany (13):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Frankfurt
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Schwerin
- Hungary (9):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gödöllő
  - Research Site, Komló
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Szigetszentmiklós
  - Research Site, Szombathely
- Israel (3):
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Rehovot
- Poland (12):
  - Research Site, Bialystok
  - Research Site, Częstochowa
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Inowrocław
  - Research Site, Katowice
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Pabianice
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zabrze
- Spain (3):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Lleida
- Ukraine (8):
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Sumy
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zhytomyr
- United Kingdom (7):
  - Research Site, Birmingham
  - Research Site, Cardiff
  - Research Site, Chorley
  - Research Site, Glasgow
  - Research Site, Hexham
  - Research Site, Liverpool
  - Research Site, Manchester

REFERENCES:
- [Derived] Sethi S, Kerwin E, Watz H, Ferguson GT, Mroz RM, Segarra R, Molins E, Jarreta D, Garcia Gil E. AMPLIFY: a randomized, Phase III study evaluating the efficacy and safety of aclidinium/formoterol vs monocomponents and tiotropium in patients with moderate-to-very severe symptomatic COPD. Int J Chron Obstruct Pulmon Dis. 2019 Mar 22;14:667-682. doi: 10.2147/COPD.S189138. eCollection 2019. PMID 30962681
- See also: Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4098&filename=D6571C00001-Protocol-Final-redacted-06Jun2018(PdfA).pdf
- See also: SAP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4098&filename=D6571C00001-SAP-Amendment-1-Final-redacted-06Jun2018(PdfA).pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted on participants with stable chronic obstructive pulmonary disease (COPD), in 11 countries: United States (US), Germany, Poland, Hungary, Bulgaria, Ukraine, United Kingdom (UK), Czech Republic, Spain, Israel & Russia (was not finally started). First participant enrolled was 05 July 2016 & participant last visit was 08 June 2017
Pre-assignment Details: Eligible Participants signed informed consent form (ICF) & entered screening (Run-in) period (14 ± 3 days), inclusion/exclusion criteria were checked by medical & COPD history, physical examination, laboratory analysis, electrocardiogram, & COPD severity (COPD Assessment Test [CAT] & post-bronchodilator forced expiratory volume in 1 second [FEV1])
Groups:
- Aclidinium Bromide (AB)/Formoterol Fumarate (FF) 400/12 μg: Randomized participants received AB 400 μg/FF 12 μg oral inhalation powder twice daily (BID) via dry powder inhaler (DPI).
- AB 400 μg: Randomized participants received AB 400 μg oral inhalation powder BID via DPI.
- FF 12 μg: Randomized participants received FF 12 μg oral inhalation powder BID via DPI.
- Tiotropium (TIO) 18 μg: Randomized participants received TIO 18 μg oral inhalation powder in capsule BID via DPI.
Period: Overall Study
Arm/Group | Aclidinium Bromide (AB)/Formoterol Fumarate (FF) 400/12 μg | AB 400 μg | FF 12 μg | Tiotropium (TIO) 18 μg
Started (All participants in the screened population who were randomized to a treatment group in the study.) | 317 | 478 | 320 | 479
Completed Treatment and Follow-up (Participants who completed the study treatment and the study, and attend to the follow-up contact) | 279 | 405 | 267 | 403
Completed (Participants who completed the study treatment and the study) | 279 | 405 | 267 | 405
Not Completed | 38 | 73 | 53 | 74
Not completed — Adverse Event | 11 | 22 | 14 | 14
Not completed — Protocol Violation | 7 | 5 | 4 | 8
Not completed — Lost to Follow-up | 1 | 5 | 2 | 2
Not completed — Lack of Efficacy | 7 | 9 | 14 | 20
Not completed — Withdrawal by Subject | 4 | 14 | 6 | 7
Not completed — Progressive disease | 6 | 15 | 13 | 18
Not completed — Reason not mentioned | 2 | 3 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclidinium Bromide (AB)/Formoterol Fumarate (FF) 400/12 μg | AB 400 μg | FF 12 μg | Tiotropium (TIO) 18 μg | Total
Number analyzed (Participants) | 314 | 475 | 319 | 475 | 1583
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Safety analysis set: All randomized participants who took at least one dose of investigational medicinal product (IMP).
  Years | 64.4 (8.5) | 64.4 (8.1) | 64.7 (8.3) | 64.0 (8.6) | 64.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety analysis set: All randomized participants who took at least one dose of IMP.
  Participants
    Female | 121 | 171 | 129 | 199 | 620
    Male | 193 | 304 | 190 | 276 | 963
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety analysis set: All randomized participants who took at least one dose of IMP.
  Participants
    American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
    Asian | 0 | 2 | 0 | 2 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 17 | 28 | 16 | 16 | 77
    White | 297 | 444 | 303 | 457 | 1501
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 1-hour Morning Post-dose Dose Forced Expiratory Volume in 1 Second (FEV1) of AB/FF 400/12 μg Compared to AB 400 μg at Week 24
Description: To assess the bronchodilatory effect by evaluating the mean changes from baseline in FEV1 at 1 hour post-dose of AB/FF 400/12 µg compared to AB 400 μg after administration of oral inhalation powder BID via DIP to participants with COPD.
  Baseline was defined as the average of the two FEV1 values measured just prior to the administration of the first dose of investigational product (IP) at randomization Visit. If one of the two was missing, then the available one would be used as baseline value.
Time Frame: At baseline 1-hour postdose and Week 24
Population: Intention-to Treat (ITT) population: All randomized participants who took at least one dose of IP and had at least a baseline FEV1, under the ITT principle and regardless the adherence to the randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: Litres
Groups:
- AB/FF 400/12 μg: Randomized participants received orally AB 400 μg/FF 12 μg inhalation powder twice daily (BID) via dry powder inhaler (DPI).
- FF 12 μg: Randomized participants received orally FF 12 μg inhalation powder BID via DPI.
- TIO 18 μg: Edit Randomized participants received orally TIO 18 μg inhalation powder in capsule BID via DPI.
Arm/Group | AB/FF 400/12 μg | AB 400 μg | FF 12 μg | TIO 18 μg
Number analyzed (Participants) | 314 | 475 | 319 | 475
Litres | 0.253 (0.013) | 0.169 (0.011) | 0.168 (0.013) | 0.161 (0.011)
Statistical Analysis 1: Comparison: AB/FF 400/12 μg vs AB 400 μg; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; LS mean difference = 0.084, 95% CI 2-sided [0.051 to 0.117]

2. Primary Outcome: Change From Baseline in Morning Predose (Trough) FEV1 of AB/FF 400/12 μg Compared to FF 12 μg at Week 24
Description: To assess the bronchodilatory effect by evaluating the mean changes from baseline in FEV1 in morning pre-dose (trough) of AB/FF 400/12 µg compared to FF 12 μg after administration of oral inhalation powder BID via DPI to participants with COPD.
  Morning pre-dose (trough) FEV1 was defined as the average of the corresponding -30 minute and 0 minute before the morning study medication at Week 24. If one time-point was missing then the available one would be used as morning pre-dose.
Time Frame: At baseline morning predose and Week 24
Population: ITT population: All randomized participants who took at least one dose of IP and had at least a baseline FEV1, under the ITT principle and regardless the adherence to the randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | AB/FF 400/12 μg | AB 400 μg | FF 12 μg | TIO 18 μg
Number analyzed (Participants) | 314 | 475 | 319 | 475
Litres | 0.080 (0.014) | 0.066 (0.012) | 0.025 (0.014) | 0.060 (0.012)
Statistical Analysis 1: Comparison: AB/FF 400/12 μg vs FF 12 μg; Test type: Superiority; p = 0.0009, Mixed model for repeated measures; LS mean difference = 0.055, 95% CI 2-sided [0.023 to 0.088]

3. Primary Outcome: Change From Baseline in Morning Predose (Trough) FEV1 at Week 24 Comparing AB 400 μg Versus TIO 18 μg to Demonstrate Non-inferiority
Description: To assess the non-inferior bronchodilatory effect by evaluating the mean changes from baseline in FEV1 in morning pre-dose (trough)of AB 400 µg compared to TIO 18 μg after administration of oral inhalation powder BID via DPI to participants with COPD.
Time Frame: At baseline morning predose and Week 24
Population: Per-Protocol (PP) population: A subset of the ITT population, consisted of participants who met all inclusion/exclusion criteria liable to affect the efficacy assessment, had sufficient treatment compliance, and did not present serious deviations of the protocol that might affect efficacy.
Measure: Least Squares Mean (Standard Error); unit: Litres
Groups:
- AB 400 μg: Randomized participants received orally AB 400 μg/FF 12 μg inhalation powder twice daily (BID) via dry powder inhaler (DPI).
- TIO 18 μg: Randomized participants received orally TIO 18 μg inhalation powder in capsule BID via DPI.
Arm/Group | AB 400 μg | TIO 18 μg
Number analyzed (Participants) | 423 | 419
Litres | 0.064 (0.013) | 0.057 (0.013)
Statistical Analysis 1: Comparison: AB 400 μg vs TIO 18 μg; Test type: Non-Inferiority — Non-inferiority was established by showing that the lower bound of the two-sided 95% confidence interval for change from baseline in morning pre-dose (trough) FEV1 at week 24 when compared AB 400 μg versus TIO 18 μg was higher than -50 mL (non-inferiority limit); p = 0.6377, Mixed model for repeated measures; LS mean difference = 0.007, 95% CI 2-sided [-0.021 to 0.035]

4. Secondary Outcome: Change From Baseline in Normalized Area Under Curve 3hours Post-dose (nAUC0-3/3h) FEV1 of AB/FF 400/12 μg Compared to AB 400 μg and and FF 12 μg at Week 24
Description: To assess the bronchodilatory effect by evaluating the mean changes from baseline in nAUC0-3/3h FEV1 of AB/FF 400/12 µg compared to AB 400 μg and and FF 12 μg after administration of oral inhalation powder BID via DPI to participants with COPD.
Time Frame: At Day 1 and Day 169
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | AB/FF 400/12 μg | AB 400 μg | FF 12 μg | TIO 18 μg
Number analyzed (Participants) | 314 | 475 | 319 | 475
Litres | 0.237 (0.013) | 0.162 (0.010) | 0.149 (0.013) | 0.151 (0.010)
Statistical Analysis 1: Comparison: AB/FF 400/12 μg vs AB 400 μg; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; LS mean difference = 0.075, 95% CI 2-sided [0.043 to 0.107]
Statistical Analysis 2: Comparison: AB/FF 400/12 μg vs FF 12 μg; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; LS mean difference = 0.087, 95% CI 2-sided [0.052 to 0.122]

5. Secondary Outcome: Responder (Number of Participants) Analysis of St. George's Respiratory Questionnaire (SGRQ) Total Score With AB/FF 400/12 μg Versus AB 400 μg and FF 12 μg.
Description: SGRQ was a A standardized self-completed tool used to measure impaired health and perceived well-being ("quality of life") in respiratory diseases. The questionnaire contained 50 items divided into 3 (symptoms, activity and impacts) dimensions. Each of the three dimensions of the questionnaire is scored separately in the range from 0 to 100%, zero score indicating no impairment of life quality. A summary score utilizing responses to all items is the total SGRQ score which also ranges from 0 to 100%. The SGRQ scores are calculated using weights attached to each item of the questionnaire which provides an estimate of the distress associated with the symptoms or state described in each item. Higher scores indicate poorer health. A decrease of at least 4 units in the SGRQ total score has been established as the criterion for minimal meaningful improvement. SGRQ responders will be those with a decrease in SGRQ total score of at least 4 units from baseline.
Time Frame: At baseline and Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AB/FF 400/12 μg | AB 400 μg | FF 12 μg | TIO 18 μg
Number analyzed (Participants) | 270 | 383 | 258 | 389
Participants
  Number of responders -Yes | 130 | 188 | 128 | 197
  Number of responders- NO | 140 | 195 | 130 | 192
Statistical Analysis 1: Comparison: AB/FF 400/12 μg vs AB 400 μg; Test type: Superiority; p = 0.8714, Logistic random-effect model; Odds ratio = 0.96, 95% CI 2-sided [0.61 to 1.51]
Statistical Analysis 2: Comparison: AB/FF 400/12 μg vs FF 12 μg; Test type: Superiority; p = 0.8873, Logistic random-effect model; Odds ratio = 0.97, 95% CI 2-sided [0.59 to 1.58]

ADVERSE EVENTS:
Time Frame: From time of signature of the ICF throughout the treatment period and including the follow-up period (14 days after the last study drug administration)
Description: An adverse event was the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition might be symptoms, signs or the abnormal results of an investigation. The safety population was defined as all randomized patients who took at least one dose of IMP.
Arm/Group | AB/FF 400/12 μg | AB 400 μg | FF 12 μg | TIO 18 μg
All-Cause Mortality (participants affected / at risk) | 1/314 | 1/475 | 4/319 | 2/475
Serious Adverse Events (participants affected / at risk) | 23/314 | 41/475 | 22/319 | 37/475
Other Adverse Events (participants affected / at risk) | 173/314 | 222/475 | 178/319 | 241/475
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AB/FF 400/12 μg (N=314) | AB 400 μg (N=475) | FF 12 μg (N=319) | TIO 18 μg (N=475)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 11 (11) | 10 (10) | 14 (14)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cor pulmonale chronic (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacunar stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AB/FF 400/12 μg (N=314) | AB 400 μg (N=475) | FF 12 μg (N=319) | TIO 18 μg (N=475)
Chronic obstructive pulmonary (Respiratory, thoracic and mediastinal disorders) | 49 (60) | 79 (90) | 58 (74) | 61 (70)
Nasopharyngitis (Infections and infestations) | 36 (42) | 47 (56) | 39 (45) | 64 (67)
Headache (Nervous system disorders) | 16 (27) | 19 (20) | 17 (19) | 25 (31)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 13 (15) | 7 (7) | 17 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 13 (18) | 6 (7) | 12 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (22) | 7 (7) | 8 (12) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 7 (7) | 4 (4) | 17 (19)
Sinusitis (Infections and infestations) | 8 (8) | 10 (10) | 6 (6) | 7 (7)
Hypertension (Vascular disorders) | 7 (7) | 8 (8) | 9 (10) | 7 (9)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1) | 6 (6) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 9 (9) | 7 (7) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 4 (4) | 3 (4) | 8 (10)
Urinary tract infection (Infections and infestations) | 4 (4) | 5 (5) | 8 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-03-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT02796677/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT02796677/SAP_001.pdf